CLINICAL TRIAL: NCT05493540
Title: Oral Ibuprofen Versus Placebo in Management of Patent Ductus Arteriosus in Preterm Infants: A Double Blind, Randomized Control Trial
Brief Title: Oral Ibuprofen Versus Placebo in Treatment of Patent Ductus Arteriosus (PDA)in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nada Youssef (Other)
Responsible Party: Sponsor-Investigator, Nada Youssef, Assistant lecturer of pediatrics and neonatology, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD 96 2020
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Patent Ductus Arteriosus After Premature Birth; Patent Ductus Arteriosus Conservative Management
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical treatment Group (Active Comparator): 40 preterm neonates will receive Ibuprofen oral suspension
  Interventions: Drug: Ibuprofen oral suspension
- Placebo Group (Placebo Comparator): 40 preterm neonates will receive oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen oral suspension — The medical treatment group will receive oral Ibuprofen with conservative therapy in the form of fluid restriction, Positive End Expiratory Pressure (PEEP), and/or diuretics
  An additional course of Ibuprofen may be offered if there is:
  1. Moderate/Severe PDA on Echocardiography
  2. Prolonged ventilation or Increased ventilatory setting
  3. Prolonged use of inotropes or vasopressors or escalating dose
     * Another form of treatment may be offered if the patient developed side effects from Ibuprofen
  Other Names: Active treatment
  Arms: Medical treatment Group
Drug: Placebo — Placebo Group will receive Oral Placebo and Conservative therapy in the form of fluid restriction, PEEP, and/or diuretics
  An Open-label option might be offered if there are concerns by attending physicians over the poor patient condition that might be attributed to persistent PDA:
  1. Prolonged Ventilation or Escalating Ventilatory Setting
  2. Prolonged Use Of Inotropes or Vasopressors or escalation of Doses
  Rescue therapy in the form of a course of oral ibuprofen may be offered:
  1. After 5 days of recruitment
  2. Moderate/Severe PDA on Echocardiography
  3. Prolonged ventilation or Increased ventilatory setting
  4. Prolonged use of inotropes or vasopressors or escalating dose - Another form of treatment may be offered if the patient developed side effects from Ibuprofen
  Other Names: Conservative
  Arms: Placebo Group

SUMMARY:
The management options of Patent Ductus Arteriosus are still controversial and differ between centers. Recently, conservative management has been gaining interest as the evidence of benefit from medical treatment in terms of mortality and morbidity is lacking.

This study will compare oral ibuprofen (the standard treatment) with the conservative treatment, in terms of ductal closure and morbidity and mortality at discharge in preterm neonates less than 34 weeks.

DETAILED DESCRIPTION:
A double-blinded, randomized, placebo-control non-inferiority trial was conducted in the neonatal intensive care unit (NICU) of Ain Shams University children's hospital, Cairo, Egypt.

Informed consent was taken from the parents or legal guardians before enrolment, after fully explaining to them the nature of the study. The approval of the Research Ethics Committee at Ain Shams University was also obtained.

All preterm neonates less than 34 weeks were assessed in the first 48 hours by clinical and echocardiographic examination by a cardiologist to detect PDA and exclude any congenital heart disease.

All neonates meeting the inclusion criteria will be randomized into one of two groups:

Medical treatment group and Placebo group. Targeted neonatal Echo was repeated after 5 days of the start of medical treatment by a neonatologist or a cardiologist to assess PDA closure.

After 7 days of intervention, open-label is offered to all patients with the option of another course for patients in the medical treatment group and Rescue therapy in the Placebo group.

The short-term morbidity is documented.

Withdrawal and replacement of individual subjects:

* The attending physician can decide to withdraw a subject from the study for urgent medical reasons. If they wish, parents or caregivers can leave the study at any time for any reason.
* Infants who are withdrawn from the study will be managed according to NICU Protocols.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 34 weeks
* PDA Size > 1.5 mm and predominantly left-to-right shunt
* One of the following:
* Signs of Pulmonary overflow: Left atrium/Aortic diameter ratio (LA/Ao), Left Ventricular End Diastolic Diameter (LVEDD).
* Signs of Systemic Hypo perfusion: Absent or Reversed diastolic flow in the aorta, celiac/mesenteric, or Anterior Cerebral Artery (ACA)/ Middle Cerebral Artery (MCA)

Exclusion Criteria:

* Chromosomal anomaly
* Congenital heart defect, other than PDA and/or patent foramen ovale
* Congenital or acquired gastrointestinal anomaly
* Previous episodes of Necrotizing enterocolitis (NEC) or intestinal perforation
* Active bleeding, especially intracranial or gastrointestinal hemorrhage
* Contraindications to the use of ibuprofen

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of PDA Closure by Echocardiography | Hospital discharge (approximately 3 months unless death occurs first)
  Compare the incidence of PDA closure assessed by Echocardiography during hospitalization between the two groups

SECONDARY OUTCOMES:
Incidence of death during hospitalization | Hospital discharge (approximately 3 months unless death occurs first)
  Compare the incidence of death during hospitalization between the two groups
Incidence of Necrotizing Enterocolitis (NEC) | Hospital discharge (approximately 3 months unless death occurs first)
  Compare the incidence of NEC during hospitalization between the two groups by Bell's staging
Incidence of Bronchopulmonary dysplasia (BPD) | Hospital discharge (approximately 3 months unless death occurs first)
  Compare the Incidence of BPD (needing supplemental oxygen at 28 days of life) during hospitalization between the two groups
Incidence of Sepsis | Hospital discharge (approximately 3 months unless death occurs first)
  Compare the Incidence of sepsis during hospitalization between the two groups by positive blood culture.
Incidence of Intraventricular hemorrhage (IVH) | Hospital discharge (approximately 3 months unless death occurs first)
  Compare the Incidence of IVH during hospitalization between the two groups by transcranial ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Nada H Youssef, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt